CLINICAL TRIAL: NCT03366025
Title: Progesterone Variation on the Final Day of Oocyte Maturation. A Prospective Cohort Study With Repeated Measurements
Brief Title: Progesterone Variation on the Final Day of Oocyte Maturation.
Status: Completed | Type: Observational
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Nikolaos Polyzos, MD PhD, Fundacion Dexeus
Other Study IDs: SMD-VPD-2017-03
Record Dates: First submitted 2017-11-28; First posted 2017-12-08 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Controlled Ovarian Stimulation; Progesterone Variation on Trigger Day; Circadian Rhythm; Oocyte Donors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oocyte donors: Healthy oocyte donors undergoing ovarian stimulation with recombinant Follicular stimulating hormone
  Interventions: Diagnostic Test: Serum progesterone measure

INTERVENTIONS:
Diagnostic Test: Serum progesterone measure — Serum Progesterone will be measured in all donors on the day triggering at 8:00 am, 12:00 p, 16:00 pm and 20:00 pm

SUMMARY:
The current study, aims through a robust design to provide a simple answer on whether progesterone levels of the same individual may significantly vary depending on the time of blood retrieval before the ovulation triggering, by evaluating the daily variability of serum progesterone on the day of triggering in healthy women who perform a COS for oocyte donation, through multiple blood samplings.

ELIGIBILITY:
Inclusion Criteria:

* Healthy oocyte donors according to spanish law for oocyte donation
* Controlled ovarian stimulation following a flexible antagonist protocol and stimulation with recombinant Follicular stimulating hormone.
* Informed consent signed

Exclusion Criteria:

* Detection of luteinizing hormone surge before triggering

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy oocyte donors according to spanish law for oocyte donation
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
Progesterone variation among 4 different moments on the day of ovulation triggering | Progesterone will be measured 4 times on the day of ovulation triggering, each of them separated 4 hours from the previous one (total 4 samples within 12 hours): blood samples will be obtained at 8:00 am, 12:00 pm, 4:00 pm and 08:00 pm
  Measurement of serum Progesterone (ng/ml) in each oocyte donor at 4 different times on the day of ovulation triggering: The primary outcome will be the variation among the 4 progesterone measurements for each patient within the fixed12 hours time (8:00am; 12:00pm; 4:00pm and 8:00pm).

CONTACTS AND LOCATIONS:
Locations (1):
- Salud de la Mujer Dexeus, Barcelona, Spain

REFERENCES:
- [Derived] Gonzalez-Foruria I, Rodriguez I, Martinez F, Rodriguez-Purata J, Montoya P, Rodriguez D, Nicolau J, Coroleu B, Barri PN, Polyzos NP. Clinically significant intra-day variability of serum progesterone levels during the final day of oocyte maturation: a prospective study with repeated measurements. Hum Reprod. 2019 Aug 1;34(8):1551-1558. doi: 10.1093/humrep/dez091. PMID 31334546